CLINICAL TRIAL: NCT03650036
Title: Pulp Therapy in Necrotic Primary Molars Using CTZ Paste and Zinc Oxide-Eugenol Paste - a Randomized Controlled Clinical Trial
Brief Title: Root Canal Treatment in Primary Molars With Necrotic Pulp Using Two Different Pulp Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Piaui (Other)
Responsible Party: Principal Investigator, Lucia de Fatima Almeida de Deus Moura, Full professor at Federal University of Piaui Dentistry course, Federal University of Piaui
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ppgo2018
Record Dates: First submitted 2018-08-18; First posted 2018-08-28 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Dental Pulp Necrosis
Keywords: Primary teeth; Dental Pulp Necrosis; Root Canal Obturation
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Endodontics

STUDY DESIGN:
Intervention Model Description: The patients will be allocated into two groups and will remain in the group until the end of the experiment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The clinical evaluations will be performed by two Paediatric Dentists who will not participate in the clinical part and will not know which group the teeth belong to. Participants also will not know in which group they will be allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): In group 1, Pulp Therapy will be done with the CTZ paste (composed of 62.5 mg of chloramphenicol, 62.5 mg of tetracycline, 125 mg of zinc oxide) will be manipulate with 0.1ml of eugenol in a sterile glass plate with flexible metal spatula at the time of use and will be taken at the tip of a number 5 exploratory probe and dispensed at the entrances of the root canals where it will be accommodated with light pressure of sterile cotton balls. The CTZ paste will be protected with a thin layer of gutta-percha, previously heated in an alcohol lamp and placed in a thin layer on the CTZ pulp. The gutta-percha blade will be condensed with medium size amalgam presser and has the objective of physically isolating the CTZ paste from the restorative material.
  Interventions: Drug: Pulp Therapy CTZ Paste
- Group 2 (Experimental): In Group 2, Pulp Therapy will be done with ZOE paste. The mechanical preparation of the root canals with 2% chlorhexidine solution and first-series K files will be performed. The instrumentation limit shall be 1 mm short of the radiographic apex. After finishing the chemical-mechanical preparation, drying of the root canals with sterile absorbent paper cones and ZOE paste insertion with K files will be performed. The zinc oxide of the ZOE paste will be supplied in 250mg capsules and handled with 0.1ml eugenol in a sterile glass plate with metal spatula at the time of use. The protection of the ZOE paste will follow the same sequence as the CTZ paste.
  Interventions: Drug: Pulp Therapy ZOE Paste

INTERVENTIONS:
Drug: Pulp Therapy CTZ Paste — CTZ paste is composed of 62.5 mg of chloramphenicol, 62.5 mg of tetracycline and 125 mg of zinc oxide and manipulated with 0.1ml of eugenol in a sterile glass plate with flexible metal spatula at the time of use.
  Other Names: Endodontic Treatment
  Arms: Group 1
Drug: Pulp Therapy ZOE Paste — The zinc oxide of the ZOE paste will be supplied in 250mg capsules and handled with 0.1ml eugenol in a sterile glass plate with metal spatula at the time of use.
  Other Names: Endodontic Treatment
  Arms: Group 2

SUMMARY:
This is a controlled, randomized, double-blind clinical study (researcher and research participant does not know which group they belong to), with the objective of evaluating clinical and radiographic performances of primary molar canal treatments with necrotic pulps using two obturator pulps. The CTZ paste (composed of chloramphenicol, tetracycline, zinc oxide and eugenol) and the ZOE paste (composed of zinc oxide and eugenol). The CTZ paste represents an alternative treatment that makes possible to treat canals of primary molars in a simplified way, without instrumentation of root canals. Studies with the CTZ pulp have demonstrated satisfactory clinical and radiographic results in addition to biocompatibility and good antimicrobial action. The zinc oxide and eugenol paste has been studied, presents good clinical and radiographic results, it is indicated by the American Academy of Paediatric Dentistry and requires mechanical chemical preparation of the root canals.

Children of both sexes, frequenters of the paediatric dentistry clinic of the Federal University of Piaui who present lower deciduous molars with clinical history and / or radiographic evidences of pulp necrosis will participate in the study.

The hypothesis of the study is that both pastes present similar clinical and radiographic results.

DETAILED DESCRIPTION:
The project followed the protocol of the Consort Statement and was approved by the Research Ethics Committee of the Federal University of Piaui ( 2,600,321) and registered in the Brazilian Registry of Clinical Trials. Software was used to determine the sample calculation that resulted in 36 teeth for each group. To minimize possible losses, the sample was increased by 20%, totalizing 86 teeth (43 per group). The teeth will be randomly allocated to two groups according to the type of pulp therapy to be used. Group 1: CTZ paste and Group 2: ZOE paste. Patients will be evaluated every three months until the end of the project, estimated at 36 months. Randomization will be performed per tooth who will receive a four-digit code, generated by Random Allocation Software, which will be present in all files of the patient, to ensure blinding of both patient and researcher. An independent individual will perform randomization, also through the same program. Numbered, opaque, and sealed sequential envelopes will be used to ensure concealment of randomization. The procedures will be performed by two researchers who will be calibrated by a researcher with experience in studies on Pulpal Therapy in primary teeth and the inter and intra-examiner concordances should be equal to or greater than 0.8, determined by the Kappa Index. A pilot study will be conducted with nine primary molars (10% of the sample) of children who will not be part of the study, to adapt the proposed methodology. Before the beginning of the pulp therapies the following protocol will be adopted: Initial radiography with infant positioners and manual processing. Guidelines for parents and children about the health/disease process, development of dental biofilm, prophylaxis with prophylactic paste, local anesthesia of inferior alveolar nerve block with 1% lidocaine with vasoconstrictor, absolute isolation of the operative field with rubber dam that will be disinfected with 2% chlorhexidine solution, tissue removal, removal of the ceiling of the pulp chamber with number 330 carbide drills spinning at high speed and under irrigation with saline solution sterile 0.9%. Afterwards, abundant washing of the pulp chamber with 2% chlorhexidine solution will be performed. Pulp therapy will follow specific protocols indicated for each group.

In group 1 (CTZ paste), the root canal entries will be located and unobstructed with the exploratory probe tip number 5, washing with 2% chlorhexidine solution, drying of the pulp chamber with sterile cotton balls, manipulation of 250 mg of the CTZ paste (composed of 62.5 mg of chloramphenicol, 62.5 mg of tetracycline, 125 mg of zinc oxide) with 0.1ml of eugenol in a sterile glass plate with flexible metal spatula at the time of use. The CTZ paste will be taken at the tip of a number 5 exploratory probe and dispensed at the entrances of the root canals where it will be accommodated with light pressure of sterile cotton balls. The CTZ paste will be protected with a thin layer of gutta-percha, previously heated in an alcohol lamp and placed in a thin layer on the CTZ pulp. The gutta-percha blade will be condensed with medium size amalgam presser and has the objective of physically isolating the CTZ paste from the restorative material.

In group 2 (ZOE paste) mechanical preparation of the root canals with 2% chlorhexidine solution and first-series K files will be performed. The instrumentation limit shall be 1 mm short of the radiographic apex. After finishing the chemical-mechanical preparation, drying of the root canals with sterile absorbent paper cones and ZOE paste insertion with K files will be performed. The zinc oxide of the ZOE paste will be supplied in 250mg capsules and handled with 0.1ml eugenol in a sterile glass plate with metal spatula at the time of use. The protection of the ZOE paste will follow the same sequence as the CTZ folder.

The teeth of both groups will be restored with high viscosity glass ionomer cement following the manufacturer 's specifications and adapted stainless steel crowns. For cementation of the steel crowns will be used glass ionomer cement for cementation following the manufacturer's specifications.

After the pulp therapies have been completed, periapical radiographs will be performed obeying the same standardization of the initial radiographs. Those responsible for the children should contact the researchers in case of any postoperative complications. Patients will be evaluated clinically and radiographically every three months until the end of the project, estimated at 36 months.

The clinical evaluations will be performed by two Paediatric Dentists who will not participate in the clinical part and will not know which group the teeth belong to and if there is a discrepancy in the evaluations, a third evaluator will be called. Radiographic evaluations will be performed by two Dental Radiologists, who will not participate in the clinical part of the study either.

The data will be entered and analysed in the Statistical Package for Social Science (SPSS® for Windows, version 22.0, SPSS Inc., Chicago, USA). Pearson's Chi-square test with the P value set at 0.05 will be performed to evaluate the results.

ELIGIBILITY:
Inclusion Criteria:

* Lower primary molars with clinical and / or radiographic history of pulp necrosis.
* Crown with sufficient dental structure to be restored with stainless steel crown.
* Rhizolysis equal to or less than 1/3.

Exclusion Criteria:

* Teeth that present calcium metamorphosis.
* Pathological root resorption.
* Coronary destruction that makes it impossible for the tooth to be restored.
* You have been using antibiotics for the last three months.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Infection control of deciduous molars with necrotic pulp by clinical examination | up to 36 months
  The methods used to evaluate the primary outcome involved clinical evaluation. Clinical evaluation will be carried out by two Pediatric Dentists who did not participate in the project and blind to which group the teeth belong to and if there is a discrepancy in evaluations, a third evaluator will be called. When there are absences of reports of pain, abscess and mobility incompatible with chronological age at the times evaluated will be considered clinical success.
Infection control of deciduous molars with necrotic pulp by Radiographic examination | up to 36 months
  The methods used to evaluate the primary outcome involved radiographic evaluation. Radiographic evaluations will be performed by two Dental Radiologists, who did not participate in the study. Radiographic success will be evidenced by the regression or absence of radiolucency in the interradicular region and absence of pathological root resorptions.

SECONDARY OUTCOMES:
1. The improvement in the Quality of life of children after pulp therapy using a questionnaire | Three months after pulp therapy.
  The Brazilian version of the Early Childhood Oral Health Impact Scale (B-ECOHIS) will be applicated for parents of children with pulp necrosis before and after pulp therapy for evaluate quality of life these children and their families after execution of the treatment. The ECOHIS consists of 13 questions divided into two main parts: child impact section (part one) and family impact section (part two). The child impact section comprises of four subscales: child symptom, child function, child psychology and child self-image/social interaction. The family impact section contains two subscales: parental distress and family function. The questionnaire is scored using a simple five-point Likert scale with responses ranging from "never" to "very often" (equivalent to a score of 0 and 4, respectively). A total score ranging from zero to 52 is calculated as a simple sum of the responses with higher scores denoting a greater oral health impact and/or poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lúcia Moura, Professor, Principal Investigator — Federal University of Piaui
Locations (1):
- Federal University of Piaui, Teresina, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No